CLINICAL TRIAL: NCT01545947
Title: A PHASE 1B, MULTI-CENTER, OPEN-LABEL STUDY OF THE MTOR KINASE INHIBITOR CC-223 IN COMBINATION WITH ERLOTINIB OR ORAL AZACITIDINE IN ADVANCED NON-SMALL CELL LUNG CANCER
Brief Title: Study Assessing Safety, Pharmacokinetics and Efficacy of CC-223 With Either Erlotinib or Oral Azacitidine in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-223-NSCL-001; 2011-005290-23 (EudraCT Number)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer
Keywords: Neoplasms; Pulmonary; Lung Cancer; Cancer of the Lung; Stage IIIB Non-Small Cell Lung Cancer; IV Non-Small Cell Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — CC-223; Erlotinib Hydrochloride; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CC-223/erlotinib concurrent (Experimental): Cohorts will receive escalating continuous daily doses (15 mg and 30 mg) of CC-223 in capsules concurrently with at least two different daily dose levels of erlotinib tablets (100 mg and 150 mg) in 28-day cycles.
  Interventions: Drug: CC-223, erlotinib
- CC-223/oral azacitidine concurrent (Experimental): Cohorts will receive escalating continuous daily doses of CC-223 (15 mg and 30 mg) with one or more dose levels of oral azacitidine (200 mg or 300 mg, as two or three 100 mg tablets) administered on Day 1 to 21 of each 28-day cycle.
  Interventions: Drug: CC-223, oral azacitidine
- CC-223/oral azacitidine sequential (Experimental): Cohorts will receive escalating continuous daily dose levels of CC-223 (15 mg and 30 mg) administered on Days 8 through 28 sequentially with one or more dose levels of of oral azacitidine (200 mg or 300 mg, as two or three 100 mg tablets) administered on Days 1 to 7 of each 28-day cycle
  Interventions: Drug: CC-223, oral azacitidine

INTERVENTIONS:
Drug: CC-223, erlotinib — Dose escalation: Combination doses start with 15 mg CC-223 and 100 mg erlotinib, or 15 mg CC-223 and 150 mg erlotonib, administered in 28-day cycles. Combination dose levels increase sequentially using predefined regimens until non-tolerated dose levels are established and a maximum tolerated dose combination has been identified for further study.
  Dose expansion: The maximum tolerated doses are evaluated further for evidence of preliminary efficacy
  Arms: CC-223/erlotinib concurrent
Drug: CC-223, oral azacitidine — Dose escalation: Combination doses start with 15 mg CC-223 and 200 mg oral azacitidine, administered in 28-day cycle. Combination dose levels increase sequentially using predefined regimens until non-tolerated dose levels are established and a maximum tolerated dose combination has been identified for further study.
  Dose expansion: The maximum tolerated doses are evaluated further for evidence of preliminary efficacy
  Arms: CC-223/oral azacitidine concurrent
Drug: CC-223, oral azacitidine — Dose escalation: Sequential dosing starts with 200 mg of oral azacitidine administered on Days 1 through 7 of each 28-day cycle, followed by daily dose level of 15 mg CC-223 on Days 8 through 28. Combination dose levels increase sequentially using predefined regimens until non-tolerated dose levels are established and a maximum tolerated dose combination has been identified for further study.
  Dose expansion: The maximum tolerated doses are evaluated further for evidence of preliminary efficacy
  Arms: CC-223/oral azacitidine sequential

SUMMARY:
The main purpose of this first study combining an investigational dual mTOR inhibitor, CC-223, with other agents (erlotinib or the investigational agent, oral azacitidine) is to establish a maximum tolerated dose level for each combination in order to evaluate their effects in future clinical trials for advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18 years or older, with histologically or cytologically-confirmed, Stage IIIB/IV Non-Small Cell Lung Cancer with tumor progression following at least one prior treatment regimen (either chemotherapy or an Epidermal Growth Factor Receptor inhibitor) for advanced disease. There is no restriction on the number of prior treatment regimens allowed.
2. Eastern Cooperative Oncology Group Performance Score of 0 to 1.
3. Adequate organ function.
4. Adequate contraception (if appropriate).
5. Consent to retrieve archival tumor tissue.
6. Consent to repeated tumor biopsy (dose expansion phase).

Exclusion Criteria:

1. Prior systemic cancer-directed treatments or investigational drugs within 4 weeks or 5 half lives, whichever is shorter except erlotinib which may be continued with intervention in subjects allocated in Arm A.
2. Symptomatic central nervous system metastases.
3. Acute or chronic pancreatitis.
4. Persistent diarrhea or malabsorption > Grade 2, despite medical management.
5. Impaired cardiac function or significant cardiac disease.
6. Diabetes on active treatment, fasting blood glucose > 126 mg/dL, HbA1c > 6.5%.
7. Known Human Immunodeficiency Virus, chronic hepatitis B or C infection.
8. Prior treatment with an investigational dual TORC1/TORC2, PI3K, or Akt inhibitor. Prior treatment with rapalogs is allowed.
9. Major surgery < 2 weeks prior to starting study drugs. No specific wash out is required for radiotherapy. Subjects must have recovered from any effects of recent therapy that might confound the safety evaluation of study drug.
10. Pregnant or breastfeeding, inadequate contraception.
11. History of concurrent second malignancies requiring ongoing systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2014-12-11 (Actual); Study Completion 2014-12-11 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 24 months
  Number of participants with adverse events
MTD | Up to 24 months
  Maximum tolerated dose (MTD)
PK-Cmax | Up to 15 months
  Pk-Maximum observed concentration in plasma (Cmax)
PK-AUC | Up to 15 months
  Area under the plasma concentration-time curve (AUC)
PK-Tmax | Up to 15 months
  PK-Time to maximum concentration (Tmax)
PK-T1/2 | Up to 15 months
  PK-Terminal half-life (T1/2)
PK-CL/F | Up to 15 months
  PK-Apparent total body clearance (CL/F)
PK-Vz/F | Up to 15 months
  PK-Apparent volume of distribution (Vz/F)

SECONDARY OUTCOMES:
mTORC1 and mTORC2 pathway biomarkers | Up to 15 months.
  The effect of treatment on mTORC1 and mTORC2 pathway biomarkers in blood and tumor
CC-223 metabolite, M1 | Up to 9 months
  CC-223 metabolite, M1, will be characterized
Tumor Response Rate | Up to 24 months
  Tumor Response Rate using RECIST 1.1 (Eisenhauer, 2009)
Number of participants surviving without tumor progression | Up to 24 months
  Number of participants surviving without tumor progression

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hege, MD, Study Director — Celgene Corporation
Locations (9):
- United States (7):
  - Cedars Sinai Medical Center, Inflammatory Bowel Disease Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - NYU School of Medicine, New York, New York
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers - Medical City, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (2):
  - Vall d´Hebron University Hospital, Barcelona
  - Hospital Virgen del Rocio Servicio de Hematologia, Seville